CLINICAL TRIAL: NCT07366983
Title: Effect of Cervical Traction From Different Angles With Neural Mobilization on Nerve Root Functions in Cervical Radiculopathy Patients
Brief Title: Effect of Cervical Traction With Neural Mobilization on Nerve Root Functions in Cervical Radiculopathy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Nagy Elshafey, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nagy-Phd
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Cervical Radiculopathy; Traction; Neural Mobilization; Nerve Root Disorder
MeSH Terms: conditions — Radiculopathy | interventions — Traction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- multimodal physical therapy program and traction with neural mobilization (30 degree) head flexion (Experimental): Patients will receive multimodal physical therapy program, and 20 min mechanical traction of cervical from 30-degree head flexion combined with neural mobilization, 3 sessions per week for 6 weeks
  Interventions: Device: traction (30 degree) head flexion; Other: Deep neck flexor strengthening exercise; Other: Sub occipital Release; Other: Hold/Relax Stretch; Other: Prone Cervical Unilateral Poster anterior Mobilization
- multimodal physical therapy program and traction with neural mobilization (30 degree) side bending (Active Comparator): Patients will receive multimodal physical therapy program, and 20 min mechanical traction of cervical while head will in 30° lateral bending to the pain-free side combined with neural mobilization, 3 sessions per week for 6 weeks.
  Interventions: Other: Deep neck flexor strengthening exercise; Other: Sub occipital Release; Other: Hold/Relax Stretch; Other: Prone Cervical Unilateral Poster anterior Mobilization; Device: traction (30 degree) side bending)
- multimodal physical therapy program and traction with neural mobilization (foramen opening position) (Active Comparator): Patients will receive multimodal physical therapy program, and 20 min mechanical traction of cervical while the head will be in 30° flexion, 15° rotation toward the painful side, and 30° lateral bending toward the pain-free side combined with neural mobilization, 3 sessions per week for 6 weeks.
  Interventions: Other: Deep neck flexor strengthening exercise; Other: Sub occipital Release; Other: Hold/Relax Stretch; Other: Prone Cervical Unilateral Poster anterior Mobilization; Device: traction (foramen opening)

INTERVENTIONS:
Device: traction (30 degree) head flexion — Triton decompression system is designed to apply traction to the cervical vertebrae in patients grouped as A, B, and C. The system includes a Triton decompression traction unit and a QuikWrapTM belting system, with traction starting from specified angles (30-degree head flexion) and an initial force of 10% of the patient's body weight, increasing by 1-2 kg as needed. Each session consists of 20 minutes of intermittent traction, allowing stress management through a bursar switch. Concurrently, neural mobilization involves shoulder depression and arm abduction, leading into either sliding or gliding of the median nerve, performed over specific sets and repetitions with designated rest periods.
  Arms: multimodal physical therapy program and traction with neural mobilization (30 degree) head flexion
Other: Deep neck flexor strengthening exercise — All patients are instructed to perform a home program involving chin-in exercises from a supine position, focusing on upper cervical spine extension and flexion. Participants will move their heads backwards and then return to the starting position, ensuring slow, controlled movements while palpating their necks to relax superficial neck muscles. The exercises will be done twice a week for six weeks, with each hold lasting 10 seconds, 15-second breaks between holds, and 10-15 repetitions in total.
Other: Sub occipital Release — In a supine position with the head on a pillow, the patient is treated by a therapist seated at the head of the table. The therapist uses both hands (digits 2 to 5) to contact the base of the occiput, gently lifting the head anteriorly while allowing the dorsum of the hands to rest on the pillow. This technique involves cranial pulling as the patient's sub occipital muscles relax, with distraction maintained for up to 5 minutes as tissue slack becomes available. Once relaxation is achieved, the therapist positions the shoulder against the patient's forehead to enhance sub occipital distraction.
Other: Hold/Relax Stretch — The therapy procedure involves positioning the patient supine and performing specific movements to address shoulder and neck tension. The therapist supports the occiput and rib area while guiding the neck into forward bending and lateral flexion, combined with right or left rotation, depending on the sequence. The patient is instructed to perform isometric contractions by elevating the shoulder against resistance for 10 seconds, followed by relaxation, with additional stretches held for 10 seconds. This process is repeated three to four times and includes a home stretching program, holding stretches for 30 to 60 seconds two to three times daily.
Other: Prone Cervical Unilateral Poster anterior Mobilization — The patient is positioned prone with a pillow under their chest, and their head and neck are in a neutral position, while the therapist stands at the head. The therapist places both thumbs on the spinous process of the targeted vertebra and applies a gentle posterior to anterior force to assess pain, mobility, and end feel, gradually increasing the force for four to five repetitions.
Device: traction (foramen opening) — Triton decompression system is designed to apply traction to the cervical vertebrae in patients grouped as A, B, and C. The system includes a Triton decompression traction unit and a QuikWrapTM belting system, with traction starting from specified angles (flexion, lateral bending and rotation according to pain) and an initial force of 10% of the patient's body weight, increasing by 1-2 kg as needed. Each session consists of 20 minutes of intermittent traction, allowing stress management through a bursar switch. Concurrently, neural mobilization involves shoulder depression and arm abduction, leading into either sliding or gliding of the median nerve, performed over specific sets and repetitions with designated rest periods.
  Arms: multimodal physical therapy program and traction with neural mobilization (foramen opening position)
Device: traction (30 degree) side bending) — Triton decompression system is designed to apply traction to the cervical vertebrae in patients grouped as A, B, and C. The system includes a Triton decompression traction unit and a QuikWrapTM belting system, with traction starting from specified angles (30 degree) side bending and an initial force of 10% of the patient's body weight, increasing by 1-2 kg as needed. Each session consists of 20 minutes of intermittent traction, allowing stress management through a bursar switch. Concurrently, neural mobilization involves shoulder depression and arm abduction, leading into either sliding or gliding of the median nerve, performed over specific sets and repetitions with designated rest periods.
  Arms: multimodal physical therapy program and traction with neural mobilization (30 degree) side bending

SUMMARY:
This study will be conducted to examine

1. The efficacy of mechanical traction from decompression angles combined with neural mobilization on the H reflex of flexor carpi radialis.
2. The efficacy of mechanical traction from decompression angles combined with neural mobilization on ultrasonography changes.
3. The efficacy of mechanical traction from decompression angles with neural mobilization has a Numeric Pain Rating Scale.
4. The efficacy of mechanical traction from decompression angles combined with neural mobilization on Neck Disability Index.

DETAILED DESCRIPTION:
Cervical radiculopathy is a condition characterized by pain, sensory and motor impairments, and slowed reflexes caused by the compression of cervical nerve roots, often stemming from cervical disc herniation. The etiology includes mechanical compression and chemical irritation, commonly due to foraminal stenosis. Cervical radiculopathy pain is a combination of nociceptive and neuropathic components, with various conservative treatments available, including immobilization and physical therapy, although evidence for their efficacy is limited. Neural mobilization especially when combined with cervical traction, shows promise in alleviating nerve-related pain and enhancing treatment adaptability. Techniques involving specific joint movements can enhance foraminal dimensions, thereby affecting nerve tension and circulation. This study uniquely examines the effects of head positions on foraminal opening and clinical outcomes, including H reflex and ultrasonography changes.

ELIGIBILITY:
Inclusion Criteria:

1. The patient's age will be ranged from 30 to 45 years old for both genders.
2. The patient's with unilateral C5-6 and C6-7 (posterior lateral disc protrusion) confirmed by T 2, axial view of magnetic resonance imaging
3. The patient's symptoms more than 3 months and positive provocative test for cervical radiculopathy (Spurling's test, shoulder abduction test, neck distraction test, and upper limb tension test 1 (Median nerve).
4. Sensory, reflex, and/ or motor changes in the upper limb

Exclusion Criteria:

1. History of surgical procedures for pathologies giving rise to neck pain or carpal tunnel syndrome
2. Clinical signs or symptoms of medical "red flags" (infection, cancer, and cardiac involvement).
3. Patients with neck pain for signs and symptoms of serious pathology, including suspected arterial insufficiency, upper cervical ligamentous insufficiency, unexplained cranial nerve dysfunction, and fracture.
4. Systemic diseases such as autoimmune and metabolic diseases.
5. History of steroid injection.
6. Complete loss of sensation along the involved nerve root.
7. bilateral radiating upper extremity
8. Diabetic polyneuropathy.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
assessment of pain intensity | at baseline and after 6 weeks
  Pain intensity was evaluated using the Numeric Pain Rating Scale (NPRS), a validated self-reported measure. Participants rated their pain on an 11-point scale from 0 (no pain) to 10 (worst pain imaginable), after receiving an explanation of the scale. NPRS scores were documented at baseline and scheduled follow-ups to track pain intensity changes during the intervention, with higher scores reflecting greater pain severity.

SECONDARY OUTCOMES:
Assessment of neck functional activities | at baseline and after 6 weeks
  The Neck Disability Index is a widely recognized tool for assessing the impact of neck pain on functional activities and measuring outcomes in clinical settings. It includes 10 questions addressing pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. The Arabic version of the Neck Disability Index is a valid instrument for evaluating disabilities in neck pain patients, demonstrating high reliability with an interclass correlation of 0.96.
assessment of H reflex for the median nerve | at baseline and after 6 weeks
  Flexor carpi radialis H-reflex is measured using an electromyogram in a semi-supine position with a supinated forearm. Hair may be removed from the anterior forearm to reduce signal resistance. The motor point of the Flexor carpi radialis is identified by applying low-threshold stimuli, aiming for the maximum response at the lowest threshold. A recording electrode is positioned at this motor point, with a reference electrode on the lateral forearm and a ground electrode proximally. To elicit the H-reflex, a surface-stimulating electrode is applied along the median nerve in the antecubital fossa.
assessment of nerve root function | at baseline and after 6 weeks
  High-resolution ultrasonography will utilize a 12- to 18-MHz linear probe to assess cervical nerve roots (NR) in seated patients with lateral neck flexion. Contralateral unaffected nerve root will serve as controls. To minimize anisotropy, the transducer will be positioned at right angles and rotated to identify the minimal cross-sectional area. C7 vertebra identification will precede imaging of the anterior and posterior tubercles of C6. The transducer will be moved to capture axial views of C5, C6, and C7 nerve roots, maintaining proximity to the transverse processes at the nerve root exit points.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Horus university, Damietta, Egypt